CLINICAL TRIAL: NCT00941343
Title: Sexuality and Management of Benign Prostatic Hyperplasia With Alfuzosin
Brief Title: Benign Prostatic Hyperplasia in Taiwan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALFUS_L_01816
Record Dates: First submitted 2009-07-16; First posted 2009-07-17 (Estimated); Last update posted 2010-03-30 (Estimated); Status verified 2010-03

CONDITIONS: Prostatic Diseases
MeSH Terms: conditions — Prostatic Diseases | interventions — alfuzosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): XATRAL 10mg OD
  Interventions: Drug: Alfuzosin (XATRAL® - SL770499)

INTERVENTIONS:
Drug: Alfuzosin (XATRAL® - SL770499) — One tablet of XATRAL® 10mg OD once a day at the end of an evening meal. The tablets had to be swallowed whole without being chewed or crushed

SUMMARY:
Primary Objective:

* To assess the sexual function of Benign Prostatic Hyperplasia patients

Secondary Objective:

* To evaluate the association between Lower Urinary Tract Symptoms severity and sexual disorders
* To compare the sexual function, urinary symptoms and Quality of Life of Benign Prostatic Hyperplasia patients on XATRAL 10mg OD among the different regions
* To correlate the Male Sexual Health Questionnaire(MSHQ) and 5-item version of the International Index of Erectile Function (IIEF-5)
* To assess the onset of action of XATRAL 10mg OD
* To assess the peak urinary flow rate
* To assess the safety and the tolerability of XATRAL 10mg OD

ELIGIBILITY:
Inclusion criteria

* Male suffering from moderate to severe lower urinary tract symptoms (LUTS), suggestive of symptomatic Benign Prostatic Hyperplasia (BPH)
* Sexually active
* Sexual attempts at least once per month

Exclusion criteria

* Known history of hepatic or severe renal insufficiency
* unstable angina pectoris
* concomitant threatening-life condition
* Previous transurethral resection of the prostate (TURP)
* Had a minimally invasive procedure within 6 months prior to inclusion
* Planned prostate surgery or minimally invasive procedure during the whole study period
* Active urinary tract infection or acute prostatitis
* Neuropathic bladder
* Diagnosed prostate cancer
* Patients having received 5-reductase inhibitors or Lower Urinary Tract Symptoms (LUTS) related phytotherapy or anti-muscarinics drug for OAB or 1-blockers within 1 month prior to inclusion
* Patients receiving any treatment for erectile dysfunction within 1 month prior to inclusion
* History of postural hypotension or syncope
* Known hypersensitivity to alfuzosin
* Patients illiterate or unable to understand or to complete the questionnaires
* Patients having participated in any clinical study in the past month
* Prostate Specific Antigen (PSA)> age specific Prostate Specific Antigen value, without using prostate biopsy to rule out prostate cancer

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 362 (Actual)
Dates: Start 2006-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Male Sexual Health Questionnaire Ejaculation score (MSHQ) | At week 24

SECONDARY OUTCOMES:
MSHQ Ejaculation score | At week 14, 12 and 24
International Prostate Symptom Score (I-PSS) including quality of life index | At week 1, 4, 12 and 24
Systolic and diastolic blood pressure | At week 1, 4, 12 and 24
Heart rate | At week 1, 4, 12 and 24
Prostate Specific Antigen | At week 24

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Chang, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Taipei, Taiwan